CLINICAL TRIAL: NCT03169166
Title: The Use of GnRH Agonist Trigger for Final Follicle Maturation in Women Undergoing Assisted Reproductive Technologies: A Prospective Randomized Controlled Trial
Brief Title: The Use of GnRH Agonist Trigger for Final Follicle Maturation in Women Undergoing Assisted Reproductive Technologies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Awwad, Professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmericanUBMCGNRH
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sterility; Infertility
Keywords: GnRH agonist; In Vitro fertilization; Assisted Reproductive Technology; Follicule Maturation; Pregnancy
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repeated 3-dose GnRHa " Triptorelin" (Experimental): Triptorelin pre-filled syringes (Gonapeptyl 0.1mg; Ferring GmbH, Germany) will be administered subcutaneously in three repeated doses 12 hours apart (0.3/0.2/0.2mg) when at least three follicles 18 mm in diameter have been observed by ultrasound examination.
  Interventions: Drug: Triptorelin
- Conventional 1-dose GnRHa " Triptorelin" (No Intervention): Triptorelin pre-filled syringes will be administered subcutaneously in a single dose (0.3 mg) when at least three follicles 18 mm in diameter have been observed by ultrasound examination.

INTERVENTIONS:
Drug: Triptorelin — Triptorelin pre-filled syringes (Gonapeptyl 0.1mg; Ferring GmbH, Germany) will be administered subcutaneously in three repeated doses 12 hours apart
  Other Names: Gonapeptyl
  Arms: Repeated 3-dose GnRHa " Triptorelin"

SUMMARY:
This is a prospective comparative randomized controlled trial investigating the effect of two GnRH agonist trigger protocols on the ongoing pregnancy rate in hyper-responder women undergoing assisted reproductive technology.

DETAILED DESCRIPTION:
Follicle maturation triggering is the final differentiation process of an immature egg before fertilization, either in normal or stimulated ovarian cycles in assisted reproductive techniques. This step has traditionally been accomplished by the administration of human chorionic gonadotropin (hCG) trigger which mimics LH activity. However, hCG is a primary cause of severe ovarian hyperstimulation syndrome (OHSS) in women and appears to initiate the complex cascade that leads to the development of serious medical complications. Numerous strategies have been suggested to prevent OHSS; one of these is the administration of a gonadotropin releasing hormone (GnRH) agonist trigger instead of hCG. Despite a high safety profile, the GnRH agonist trigger of follicle maturation was found to be associated with a decreased probability of clinical and ongoing pregnancy rates and very high miscarriage rates. A profoundly deficient luteal phase is believed to be the cause of compromised reproductive outcome. Our personal clinical practice at the AUBMC Fertility Center seems to indicate that a novel GnRH agonist administration protocol is associated with a comparable reproductive performance to standard hCG trigger. In this study, we aim to validate the above clinical impression and assess associated parameters of success. Therefore, a prospective comparative randomized controlled trial will be performed in order to investigate the effect of three repeated doses of GnRH agonist trigger "Triptorelin" accompanied by intensive Luteal Support on the ongoing pregnancy outcome in women who are hyper-responders to ovarian stimulation when undergoing assisted reproductive technology.

ELIGIBILITY:
Inclusion Criteria:

* Normal uterine cavity (as assessed by hysteroscopy or HSG).
* Normal hormonal investigation: TSH, PRL.
* More than 15 follicles (≥12 mm in diameter) on ultrasound, and/or estradiol level of > 3500 pg/ml on the day of trigger.

Exclusion Criteria:

* History of three or more miscarriages.
* History of three or more previous IVF failures.
* Abnormal uterine cavity (Hysteroscopy or HSG).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 277 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate in hyper-responder women undergoing assisted reproductive technology cycles | 20 weeks from Last Menstrual Period (LMP)

SECONDARY OUTCOMES:
Oocyte collection rate | On the day of ovum pick-up
  oocyte maturation rate ovarian volume on the day of hCG titer

OTHER OUTCOMES:
Fertilization rate | 16-18 hours post insemination
Total pregnancy rate | 10-12 days from embryo transfer
Clinical pregnancy rate | 7 weeks from LMP
Implantation rate | 7 weeks from LMP
Miscarriage rate | From a positive pregnancy test till 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Awwad, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided